CLINICAL TRIAL: NCT04090177
Title: Evaluation of a Peer-led eHealth Wheelchair Skills Training Program: Training to Enhance Adaptation and Management for Wheelchair Users
Brief Title: Training to Enhance Adaptation and Management for Wheelchair Users (TEAMWheels)
Acronym: TEAMWheels
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Manitoba (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Laval University (Other); University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: #50326/321741; HS22711 (H2019:124) (Other: University of Manitoba Health Research Ethics Board)
Record Dates: First submitted 2019-09-11; First posted 2019-09-16 (Actual); Last update posted 2023-11-29 (Actual); Status verified 2023-11

CONDITIONS: Mobility Limitation
MeSH Terms: conditions — Mobility Limitation

STUDY DESIGN:
Intervention Model Description: The treatment group receives the TEAM Wheels program over a 4-week period. Three virtual/teleconference (MS Teams) sessions will be arranged between the peer-trainer and participant, about 1 week apart. Peer trainers are experienced MWC users trained to deliver the TEAM Wheels program. After Session 1, participants engage in 4 weeks of eHealth home program training. They are asked to practice for 75-150 minutes per week, in 15-30 minute blocks, 1-2 times/day, 3-5 days/week. The control group receives no intervention over the 4-wk period ("usual practice"). Control group participants placed on the wait-list will receive the TEAM Wheels program following completion of the study. Any formal MWC training received during the wait-list period will be documented for potential post-hoc analysis as a confounding variable; research evidence and clinical experience confirm that in all 3 provinces formal training is not provided once MWC users are discharged from hospital.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Neither the investigators nor the biostatistician/outcomes assessor will know the intervention arm to which study participants have been assigned. A unique study ID will be assigned to each study participant and as well as a unique code to distinguish which intervention arm to which each participant is randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention-TEAM Wheels (Experimental): The treatment group will receive the TEAM Wheels program over a 4-week period. Session 1 will be virtually delivered via MS Teams teleconference. The peer trainer is an experienced MWC user trained to deliver the TEAM Wheels program. At least 2 peers will be trained at each site to offer multiple trainer attributes; a male and female, one being at least 50 years old. Participants will pre-select a peer trainer from a biosketch to optimize training effect (e.g., preference for age, sex factors); comparability in age has been identified as preferential among older adults and influential to self-efficacy. After Session 1, participants engage in 4 weeks of eHealth home program training. They are instructed to practice for 75-150 minutes/week. Consistent with motor learning principles, we encourage training in 15-30 minute blocks 1-2 times/day, 3-5 days/week. The peer trainer arranges the remaining two virtual teleconference sessions with the participant, about 1 week apart.
  Interventions: Behavioral: TEAM Wheels
- Control-Wait List (No Intervention): The control group receives no specific intervention over the course of the 4-week period. This reflects "usual practice"/typical experience of a MWC user in their provincial context. Control group participants placed on the wait-list will receive the TEAM Wheels program following completion of the study (i.e. after post-treatment data collection). The site Research Coordinator/Assistant will make telephone or email contact with control group participants at the end of weeks 2 and 4 during the study period to deter attrition/drop-out. When contact is made at week 4, the Research Coordinator will schedule an appointment for post-treatment data collection (week 7). Any formal MWC training received during the wait-list period will be documented for potential post-hoc analysis as a confounding variable; research evidence and investigators' clinical experience confirm that in all 3 provinces formal training is not provided once MWC users are discharged from hospital.

INTERVENTIONS:
Behavioral: TEAM Wheels — A 1-month, peer-led, eHealth training program (TEAM Wheels) for individuals transitioning to manual wheelchair use to improve satisfaction with activity participation and related rehabilitation outcomes.
  Arms: Intervention-TEAM Wheels

SUMMARY:
The purpose of this study is to evaluate the effect of a 1-month, peer-led eHealth training program (TEAM Wheels) on satisfaction with activity participation and related rehabilitation outcomes among individuals transitioning to manual wheelchair use, compared with current wheelchair training practice. The primary objectives include: 1. Measuring the effect of TEAM Wheels on satisfaction with participation in important activities of life compared to current practice; 2. Measuring retention of participation benefits at 6-months post treatment. Secondary Objectives relate to additional rehabilitation Outcomes and include: 1. Comparing the effect of TEAM Wheels to current practice on wheelchair skills capacity and performance; wheelchair-specific self-efficacy; health-related quality of life; and objective measurement of wheelchair mobility. 2. Measuring retention of rehabilitation outcome benefits at 6-months post treatment.

DETAILED DESCRIPTION:
This study will use a three-site (Winnipeg, Vancouver, and Quebec City) randomized controlled trial to compare differences in current wheelchair training practice and a 1-month, peer-led (virtual due to SARS-CoV-2; COVID-19) eHealth training program (TEAM Wheels). Subjects will randomly be assigned to the TEAM Wheels or control group using a 1:1 allocation ratio between groups. To support balance between groups and masking of assignment, our statistician will create a computerized randomization process with undisclosed block size. Once subjects are enrolled, baseline data will be collected and entered into a secure database. A site coordinator or assistant will then obtain the participant's group assignment and coordinate the first in-person peer trainer session. For treatment group assignments this will occur as soon as it is practical and for control group assignments this will be scheduled after blinded post-treatment data collection is complete. To address bias, subjects will be instructed not to discuss their program.

The treatment group will receive the TEAM Wheels program over a 4-week period. An initial meeting (Session 1) will be arranged via teleconference (MS Teams). The peer trainer is an experienced Manual Wheelchair (MWC) user trained to deliver the TEAM Wheels program. At least 2 peers will be hired and trained at each site to offer multiple trainer attributes. We will intentionally include a male and female, one being at least 50 years of age. Participants will pre-select a peer trainer based on a biosketch to optimize training effect (e.g., preference for age, sex factors); comparability in age has been identified as preferential among older adults and influential to self-efficacy. Following Session 1, participants engage in 4 weeks of training with the eHealth home program. They are instructed to practice for 75 to 150 minutes per week. Consistent with motor learning principles, we encourage training in 15-30 minute blocks 1-2 times per day, 3-5 days per week. The peer trainer will arrange with the participant the remaining two virtual sessions, approximately one week apart.

Control Group. The control group receives no specific intervention over the course of the 4-week period. This reflects "usual practice" or the typical experience of a MWC user in their provincial context. Control group participants placed on the wait-list will receive the TEAM Wheels program, as described, following completion of the study (i.e. after post-treatment data collection). The site Research Coordinator will make telephone or email contact with control group participants at the end of weeks 2 and 4 during the study period to deter attrition/drop-out. When contact is made at week 4, the Research Coordinatort will schedule an appointment for post-treatment data collection (week 7). Any formal MWC training received during the wait-list period will be documented for potential post-hoc analysis as a confounding variable; however, research evidence and the investigators' clinical experience confirm that in all 3 provinces formal training is not provided once MWC users are discharged from hospital.

Assessments. The outcome measures will be collected at baseline (pre-randomization) and post-intervention. A Research Assistant/Coordinator at each site will contact the participant via MS Teams videoconference at baseline and subsequent data collection points to administer the outcome measures. Participants will be shown a video to help them apply an Actigraph device (i.e. small battery-operated accelerometer) to the participant's wheelchair spokes and after 2 weeks will either retrieve it or provide a self-addressed stamped envelope for the participant to return via post. Post-treatment data will be collected at week 7 to incorporate a 2-week window for consolidation of learning following the 4-week intervention. Follow-up (retention) data will be collected from treatment group participants 6 months later (week 31).

Outcome measures. At baseline, descriptive characteristics including age, sex, gender, marital status, the highest level of education, primary diagnoses related to MWC use, Wheel diameter, and length of time using the MWC will be collected. Five outcome measures will be administered at baseline, post-treatment, and 6-month follow-up (for treatment group participants).

Wheelchair Skills Test - Questionnaire (WST-Q). To address environmental barriers, MWC users must learn specific mobility skills such as managing inclines, thresholds, and doorways. This is of considerable importance since training also involves learning to recognize risks and limitations. WST-Q evaluates 34 discrete skills; respondents rate their capacity (i.e. ability) with each skill as well as performance frequency. Capacity is rated as Yes (2), Yes with difficulty (1), or No (0); performance is rated as Always (2), Sometimes (1), or Never (0). Total skill Capacity (0-100%) and Performance (0-100%) scores are calculated. The WST has demonstrated excellent reliability for test-retest (ICC=0.90), intra-rater (ICC=0.96), and inter-rater (ICC=0.97) administration.

Wheelchair Outcome Measure (WhOM). The rehabilitation literature strongly suggests that intervention outcomes should include not only externally defined measures but also measures of user-identified activities of relevance and perceived satisfaction with performance. A 2008 review of wheelchair-specific outcomes found the WhOM was the only tool that included activities selected and weighted by the user and featured participation in social roles.Two published literature reviews identify the WhOM as the most client-centred and psychometrically robust tool among participation outcomes for wheelchair users. WhOM is administered as a semi-structured interview. Respondents identify 10 activities (5 performed inside and 5 performed outside of the home), rating their satisfaction with performance on an 11-point scale (0-10) for each activity. The WhOM demonstrates good reliability (Test-retest ICC = 0.83-0.88; Inter-rater ICC = 0.90-0.91) and validity (correlations with LIFE-H: rs = 0.3-0.5) in use among individuals with spinal cord injury and older adults (Test-retest ICC = 0.77-1.00; correlation with QUEST rs = 0.36 -0.45).

Wheelchair Use Confidence Scale-(WheelCon-SF). Self-efficacy has been identified as a key component in the performance of wheelchair mobility skills. Incorporating the principles of cognitive theory, including self-efficacy, can promote program adherence and skill acquisition. Preliminary research has suggested that standardized training can increase wheelchair confidence among older adults. WheelCon-SF is a self-report questionnaire with 21 statements related to confidence using a wheelchair in various activities and environments. Items are rated on a scale from 0 ("not confident") to 10 ("completely confident"), providing a total mean score (0-10). The WheelCon-SF is more responsive than the original 65-item version; a recent study reported high test-retest reliability (ICC=0.98) and internal consistency (Cronbach's alpha = 0.95).

The Short-Form 36 (SF-36) Health Survey Questionnaire is a measure of health status across the following domains: physical function, physical limitations, emotional limitations, pain, social function, energy, perceived health, and mental health. The literature identifies inherent wording bias of the mobility-related SF-36 test items, which presume ambulation as a norm so we opted to use the Enabled version that explicitly acknowledges the use of a mobility aid and replaces the words "climbing" and "walking" with "going". Short Form-36E (Enabled) is specific to the study population of manual wheelchair users and will provide detailed and specific data related to HRQL.

Objective Wheelchair Mobility. To triangulate measurement of improvement in mobility and community engagement, accelerometry data (ActigraphTM, Pensacola FL) will be used to objectively measure MWC activation over a 10-day period at baseline, post-treatment, and follow-up data collection points. The Actigraph is attached to a rear wheel on the MWC; a battery provides up to 14 days of passive data collection without impeding MWC operation. Data loggers have demonstrated valid and reliable measurement of MWC movement, with accuracy beyond 90%. A tri-axial accelerometer records acceleration forces during MWC use, downloadable as a .csv file. Algorithms developed by our team convert data into total and mean values of distance, speed, and 'bout' frequency (meaningful transitions between functional activities), parameters that reflect mobility patterns and activity of MWC users which we expect to change as a result of improvements in skill and participation.

Program details TEAM Wheels is a 4-week, community-based, tailored program integrating eHealth and peer-led components to optimize learning while limiting the time demands of health care professionals. The eHealth component is a 10" computer tablet with a custom training application. The tablet mounts conveniently on the lap for "in-chair" training, enabling MWC users to learn and practice mobility skills in authentic contexts of home and community. The interactive application includes a structured curriculum with over 200 video clips featuring education, peer demonstration, and training activities. The peer-led component involves experienced MWC users with specialized training who can leverage their own experience and ability to relate as influential peers. The peer trainer conducts 3 virtual/teleconference (MS Teams) sessions with the participant, negotiating individualized goals, introducing wheelchair skills and management strategies, and providing an orientation to the eHealth home program. Peer trainers monitor eHealth training activity, which the tablet uploads to a secure website, intervening or modifying the program when required. Additional communication can be initiated between MWC user and peer trainer using a video messaging through MS Teams (on the computer tablet). The tablet is menu driven and interactive, using a touch-screen interface. A tablet offers considerable advantages over traditional paper/hand-out home programs. Training is provided in a multi-modal format with illustrations and videos, allowing detailed step-by-step guidance, close-ups, and demonstrations using age-appropriate older adult models. Practice activities can be clearly demonstrated (to ensure they are performed appropriately) and include imitative, function-based, and interactive game-related activities. Subjects can also contact their Peer-Trainer using the MS Teams (on the tablet); Trainers will review and respond within 48 hours. The tablet is housed in a rigid case with a simple strap that wraps around the participant's thighs. Subjects can secure the tablet on their lap and practice anywhere in their home or community, or place the tablet on another surface for viewing or video recording. Training activities are highlighted/checked off after completion, indicating to the subject they can advance to the next component. A "Progress" tab provides regular updates on the number of minutes practiced each week to reinforce adherence. The tablet will have Internet access for communication and data transfer/update capability, but the training program can operate in stand-alone mode as well.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* use a MWC (even part time)
* living in the community
* have the ability to propel with both arms
* have sufficient language abilities to engage with the training material in English,

Exclusion Criteria:

* have a health condition that might interfere with training (e.g., cancer; surgery)
* concurrently receiving any MWC skills training beyond that of typical practice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Satisfaction with Participation: Wheelchair Outcome Measure (WhOM) | Baseline
  WhOM has been found to be the only tool that includes activities selected and weighted by the user and featured participation in social roles. WhOM has been identified as the most client-centred and psychometrically robust tool among participation outcomes for wheelchair users. It is administered as a semi-structured interview. Respondents identify 10 activities (5 performed inside and 5 performed outside of the home), rating their satisfaction with performance on an 11-point scale (0-10) for each activity. The WhOM demonstrates good reliability (Test-retest ICC = 0.83-0.88; Inter-rater ICC = 0.90-0.91) and validity (correlations with LIFE-H: rs = 0.3-0.5) in use among individuals with spinal cord injury and older adults (Test-retest ICC = 0.77-1.00; correlation with QUEST rs = 0.36 -0.45).
Satisfaction with Participation: Wheelchair Outcome Measure (WhOM) | Post-Treatment (Week 7)
  WhOM has been found to be the only tool that includes activities selected and weighted by the user and featured participation in social roles. WhOM has been identified as the most client-centred and psychometrically robust tool among participation outcomes for wheelchair users. It is administered as a semi-structured interview. Respondents identify 10 activities (5 performed inside and 5 performed outside of the home), rating their satisfaction with performance on an 11-point scale (0-10) for each activity. The WhOM demonstrates good reliability (Test-retest ICC = 0.83-0.88; Inter-rater ICC = 0.90-0.91) and validity (correlations with LIFE-H: rs = 0.3-0.5) in use among individuals with spinal cord injury and older adults (Test-retest ICC = 0.77-1.00; correlation with QUEST rs = 0.36 -0.45).
Satisfaction with Participation: Wheelchair Outcome Measure (WhOM) | 6-Month Follow-up (Week 31)
  WhOM has been found to be the only tool that includes activities selected and weighted by the user and featured participation in social roles. WhOM has been identified as the most client-centred and psychometrically robust tool among participation outcomes for wheelchair users. It is administered as a semi-structured interview. Respondents identify 10 activities (5 performed inside and 5 performed outside of the home), rating their satisfaction with performance on an 11-point scale (0-10) for each activity. The WhOM demonstrates good reliability (Test-retest ICC = 0.83-0.88; Inter-rater ICC = 0.90-0.91) and validity (correlations with LIFE-H: rs = 0.3-0.5) in use among individuals with spinal cord injury and older adults (Test-retest ICC = 0.77-1.00; correlation with QUEST rs = 0.36 -0.45).

SECONDARY OUTCOMES:
Wheelchair Skills Test - Questionnaire (WST-Q) | Baseline
  To address environmental barriers, MWC users must learn specific mobility skills such as managing inclines, thresholds, and doorways. This is of considerable importance since training also involves learning to recognize risks and limitations. WST-Q evaluates 34 discrete skills; respondents rate their capacity (i.e. ability) with each skill as well as performance frequency. Capacity is rated as Yes (2), Yes with difficulty (1), or No (0); performance is rated as Always (2), Sometimes (1), or Never (0). Total skill Capacity (0-100%) and Performance (0-100%) scores are calculated. The WST has demonstrated excellent reliability for test-retest (ICC=0.90), intra-rater (ICC=0.96), and inter-rater (ICC=0.97) administration.
Wheelchair Skills Test - Questionnaire (WST-Q) | Post-Treatment (Week 7)
  To address environmental barriers, MWC users must learn specific mobility skills such as managing inclines, thresholds, and doorways. This is of considerable importance since training also involves learning to recognize risks and limitations. WST-Q evaluates 34 discrete skills; respondents rate their capacity (i.e. ability) with each skill as well as performance frequency. Capacity is rated as Yes (2), Yes with difficulty (1), or No (0); performance is rated as Always (2), Sometimes (1), or Never (0). Total skill Capacity (0-100%) and Performance (0-100%) scores are calculated. The WST has demonstrated excellent reliability for test-retest (ICC=0.90), intra-rater (ICC=0.96), and inter-rater (ICC=0.97) administration.
Wheelchair Skills Test - Questionnaire (WST-Q) | 6-Month Follow-up (Week 31)
  To address environmental barriers, MWC users must learn specific mobility skills such as managing inclines, thresholds, and doorways. This is of considerable importance since training also involves learning to recognize risks and limitations. WST-Q evaluates 34 discrete skills; respondents rate their capacity (i.e. ability) with each skill as well as performance frequency. Capacity is rated as Yes (2), Yes with difficulty (1), or No (0); performance is rated as Always (2), Sometimes (1), or Never (0). Total skill Capacity (0-100%) and Performance (0-100%) scores are calculated. The WST has demonstrated excellent reliability for test-retest (ICC=0.90), intra-rater (ICC=0.96), and inter-rater (ICC=0.97) administration.
Wheelchair Use Confidence Scale-(WheelCon-SF) | Baseline
  Self-efficacy has been identified as a key component in the performance of wheelchair mobility skills. Incorporating the principles of cognitive theory, including self-efficacy, can promote program adherence and skill acquisition. Preliminary research has suggested that standardized training can increase wheelchair confidence among older adults. WheelCon-SF is a self-report questionnaire with 21 statements related to confidence using a wheelchair in various activities and environments. Items are rated on a scale from 0 ("not confident") to 10 ("completely confident"), providing a total mean score (0-10).27 The WheelCon-SF is more responsive than the original 65-item version; a recent study reported high test-retest reliability (ICC=0.98) and internal consistency (Cronbach's alpha = 0.95).
Wheelchair Use Confidence Scale-(WheelCon-SF) | Post-Treatment (Week 7)
  Self-efficacy has been identified as a key component in the performance of wheelchair mobility skills. Incorporating the principles of cognitive theory, including self-efficacy, can promote program adherence and skill acquisition. Preliminary research has suggested that standardized training can increase wheelchair confidence among older adults. WheelCon-SF is a self-report questionnaire with 21 statements related to confidence using a wheelchair in various activities and environments. Items are rated on a scale from 0 ("not confident") to 10 ("completely confident"), providing a total mean score (0-10).27 The WheelCon-SF is more responsive than the original 65-item version; a recent study reported high test-retest reliability (ICC=0.98) and internal consistency (Cronbach's alpha = 0.95).
Wheelchair Use Confidence Scale-(WheelCon-SF) | 6-Month Follow-up (Week 31)
  Self-efficacy has been identified as a key component in the performance of wheelchair mobility skills. Incorporating the principles of cognitive theory, including self-efficacy, can promote program adherence and skill acquisition. Preliminary research has suggested that standardized training can increase wheelchair confidence among older adults. WheelCon-SF is a self-report questionnaire with 21 statements related to confidence using a wheelchair in various activities and environments. Items are rated on a scale from 0 ("not confident") to 10 ("completely confident"), providing a total mean score (0-10).27 The WheelCon-SF is more responsive than the original 65-item version; a recent study reported high test-retest reliability (ICC=0.98) and internal consistency (Cronbach's alpha = 0.95).
Short Form-36E (Enabled) | Baseline
  Full title: Short Form 36 Health Survey Questionnaire (SF-36) (Enabled) 'Enabled' indicates wording is included above terms requiring adaptation for individuals requiring mobility assistive devices (the word "go" replaces "walk" and "climb").
  SF-36E is a questionnaire specific to the study population of manual wheelchair users that provides detailed data related to HRQL specific to this population, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Short Form-36E (Enabled) | Post-Treatment (Week 7)
  Full title: Short Form 36 Health Survey Questionnaire (SF-36) (Enabled) 'Enabled' indicates wording is included above terms requiring adaptation for individuals requiring mobility assistive devices (the word "go" replaces "walk" and "climb").
  SF-36E is a questionnaire specific to the study population of manual wheelchair users that provides detailed data related to HRQL specific to this population, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Short Form-36E (Enabled) | 6-Month Follow-up (Week 31)
  Full title: Short Form 36 Health Survey Questionnaire (SF-36) (Enabled) 'Enabled' indicates wording is included above terms requiring adaptation for individuals requiring mobility assistive devices (the word "go" replaces "walk" and "climb").
  SF-36E is a questionnaire specific to the study population of manual wheelchair users that provides detailed data related to HRQL specific to this population, which measures eight domains of health status: physical functioning (10 items); physical role limitations (four items); bodily pain (two items); general health perceptions (five items); energy/vitality (four items); social functioning (two items); emotional role limitations (three items) and mental health (five items). A scoring algorithm is used to convert the raw scores into the eight dimensions listed above. The scores are transformed to range from zero where the respondent has the worst possible health to 100 where the respondent is in the best possible health.
Objective Wheelchair Mobility | Baseline
  To triangulate measurement of improvement in mobility and community engagement, accelerometry data (ActigraphTM, Pensacola FL) will be used to objectively measure MWC activation over a 10-day period at baseline, post-treatment, and follow-up data collection points. The Actigraph is attached to a rear wheel on the MWC; a battery provides up to 14 days of passive data collection without impeding MWC operation. Data loggers have demonstrated valid and reliable measurement of MWC movement, with accuracy beyond 90%. A tri-axial accelerometer records acceleration forces during MWC use, downloadable as a .csv file. Algorithms developed by our team convert data into total and mean values of distance, speed, and 'bout' frequency (meaningful transitions between functional activities), parameters that reflect mobility patterns and activity of MWC users which we expect to change as a result of improvements in skill and participation.
Objective Wheelchair Mobility | 2-weeks
  To triangulate measurement of improvement in mobility and community engagement, accelerometry data (ActigraphTM, Pensacola FL) will be used to objectively measure MWC activation over a 10-day period at baseline, post-treatment, and follow-up data collection points. The Actigraph is attached to a rear wheel on the MWC; a battery provides up to 14 days of passive data collection without impeding MWC operation. Data loggers have demonstrated valid and reliable measurement of MWC movement, with accuracy beyond 90%. A tri-axial accelerometer records acceleration forces during MWC use, downloadable as a .csv file. Algorithms developed by our team convert data into total and mean values of distance, speed, and 'bout' frequency (meaningful transitions between functional activities), parameters that reflect mobility patterns and activity of MWC users which we expect to change as a result of improvements in skill and participation.
Objective Wheelchair Mobility | 6-Month Follow-up
  To triangulate measurement of improvement in mobility and community engagement, accelerometry data (ActigraphTM, Pensacola FL) will be used to objectively measure MWC activation over a 10-day period at baseline, post-treatment, and follow-up data collection points. The Actigraph is attached to a rear wheel on the MWC; a battery provides up to 14 days of passive data collection without impeding MWC operation. Data loggers have demonstrated valid and reliable measurement of MWC movement, with accuracy beyond 90%. A tri-axial accelerometer records acceleration forces during MWC use, downloadable as a .csv file. Algorithms developed by our team convert data into total and mean values of distance, speed, and 'bout' frequency (meaningful transitions between functional activities), parameters that reflect mobility patterns and activity of MWC users which we expect to change as a result of improvements in skill and participation.

OTHER OUTCOMES:
Cost | Post-treatment (Week 7)
  To measure costs of the intervention in order to conduct an economic evaluation from the perspective of a health service provider. Costs include material (such as tablets, internet access for the duration of the intervention) and human resources (such as peer trainer time).

CONTACTS AND LOCATIONS:
Overall Officials: Ed Giesbrecht, PhD, Principal Investigator — University of Manitoba
Locations (3):
- Canada (3):
  - University of British Columbia, Vancouver, British Columbia
  - University of Manitoba, Winnipeg, Manitoba
  - Universite Laval, Québec

IPD SHARING:
Plan to Share IPD: Yes
Specific individual participant data sets to be shared include all collected IPD.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be made available starting six months after publication of study findings in a peer reviewed journal.
Access Criteria: Data access requests will be reviewed by the appropriate review panel. Requestors will be required to sign a Data Access/Sharing Agreement.

REFERENCES:
- [Background] Giesbrecht EM, Miller WC. A randomized control trial feasibility evaluation of an mHealth intervention for wheelchair skill training among middle-aged and older adults. PeerJ. 2017 Oct 5;5:e3879. doi: 10.7717/peerj.3879. eCollection 2017. PMID 29018615
- [Background] Best KL, Miller WC, Routhier F, Eng JJ. Feasibility of the trial procedures for a randomized controlled trial of a community-based peer-led wheelchair training program for older adults. Pilot Feasibility Stud. 2017 Jul 17;4:18. doi: 10.1186/s40814-017-0158-3. eCollection 2018. PMID 28725451
- [Background] Best KL, Miller WC, Eng JJ, Routhier F, Goldsmith C. Randomized controlled trial protocol feasibility: The Wheelchair Self-Efficacy Enhanced for Use (WheelSeeU). Can J Occup Ther. 2014 Dec;81(5):308-19. doi: 10.1177/0008417414546743. PMID 25702375
- [Background] Best KL, Miller WC, Huston G, Routhier F, Eng JJ. Pilot Study of a Peer-Led Wheelchair Training Program to Improve Self-Efficacy Using a Manual Wheelchair: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 Jan;97(1):37-44. doi: 10.1016/j.apmr.2015.08.425. Epub 2015 Sep 4. PMID 26343171
- [Background] Smith EM, Giesbrecht EM, Mortenson WB, Miller WC. Prevalence of Wheelchair and Scooter Use Among Community-Dwelling Canadians. Phys Ther. 2016 Aug;96(8):1135-42. doi: 10.2522/ptj.20150574. Epub 2016 Feb 4. PMID 26847009
- [Background] Giesbrecht EM, Smith EM, Mortenson WB, Miller WC. Needs for mobility devices, home modifications and personal assistance among Canadians with disabilities. Health Rep. 2017 Aug 16;28(8):9-15. PMID 29044443
- [Background] Shields M. Use of wheelchairs and other mobility support devices. Health Rep. 2004 May;15(3):37-41. No abstract available. PMID 15208888
- [Background] Finlayson M, van Denend T. Experiencing the loss of mobility: perspectives of older adults with MS. Disabil Rehabil. 2003 Oct 21;25(20):1168-80. doi: 10.1080/09638280310001596180. PMID 14534060
- [Background] Simpson RC, LoPresti EF, Cooper RA. How many people would benefit from a smart wheelchair? J Rehabil Res Dev. 2008;45(1):53-71. doi: 10.1682/jrrd.2007.01.0015. PMID 18566926
- [Background] Rudman DL, Hebert D, Reid D. Living in a restricted occupational world: the occupational experiences of stroke survivors who are wheelchair users and their caregivers. Can J Occup Ther. 2006 Jun;73(3):141-52. doi: 10.2182/cjot.05.0014. PMID 16871856
- [Background] Kirby RL, Ackroyd-Stolarz SA, Brown MG, Kirkland SA, MacLeod DA. Wheelchair-related accidents caused by tips and falls among noninstitutionalized users of manually propelled wheelchairs in Nova Scotia. Am J Phys Med Rehabil. 1994 Sep-Oct;73(5):319-30. doi: 10.1097/00002060-199409000-00004. PMID 7917161
- [Background] Gavin-Dreschnack D, Nelson A, Fitzgerald S, Harrow J, Sanchez-Anguiano A, Ahmed S, Powell-Cope G. Wheelchair-related falls: current evidence and directions for improved quality care. J Nurs Care Qual. 2005 Apr-Jun;20(2):119-27. doi: 10.1097/00001786-200504000-00006. PMID 15839290
- [Background] Tu CJ, Liu L, Wang W, Du HP, Wang YM, Xu YB, Li P. Effectiveness and safety of wheelchair skills training program in improving the wheelchair skills capacity: a systematic review. Clin Rehabil. 2017 Dec;31(12):1573-1582. doi: 10.1177/0269215517712043. Epub 2017 Jun 5. PMID 28580801
- [Background] Keeler L, Kirby RL, Parker K, McLean KD, Hayden JA. Effectiveness of the Wheelchair Skills Training Program: a systematic review and meta-analysis. Disabil Rehabil Assist Technol. 2019 May;14(4):391-409. doi: 10.1080/17483107.2018.1456566. Epub 2018 Apr 4. PMID 29616832
- [Background] MacPhee AH, Kirby RL, Coolen AL, Smith C, MacLeod DA, Dupuis DJ. Wheelchair skills training program: A randomized clinical trial of wheelchair users undergoing initial rehabilitation. Arch Phys Med Rehabil. 2004 Jan;85(1):41-50. doi: 10.1016/s0003-9993(03)00364-2. PMID 14970966
- [Background] Worobey LA, Kirby RL, Heinemann AW, Krobot EA, Dyson-Hudson TA, Cowan RE, Pedersen JP, Shea M, Boninger ML. Effectiveness of Group Wheelchair Skills Training for People With Spinal Cord Injury: A Randomized Controlled Trial. Arch Phys Med Rehabil. 2016 Oct;97(10):1777-1784.e3. doi: 10.1016/j.apmr.2016.04.006. Epub 2016 May 3. PMID 27153762
- [Background] Best KL, Kirby RL, Smith C, MacLeod DA. Wheelchair skills training for community-based manual wheelchair users: a randomized controlled trial. Arch Phys Med Rehabil. 2005 Dec;86(12):2316-23. doi: 10.1016/j.apmr.2005.07.300. PMID 16344029
- [Background] Ozturk A, Ucsular FD. Effectiveness of a wheelchair skills training programme for community-living users of manual wheelchairs in Turkey: a randomized controlled trial. Clin Rehabil. 2011 May;25(5):416-24. doi: 10.1177/0269215510386979. Epub 2010 Nov 8. PMID 21059666
- [Background] Kirby RL. Wheelchair skills assessment and training. Boca Raton, FL: CRC Press, Taylor & Francis Group, 2017.
- [Background] Best KL, Routhier F, Miller WC. A description of manual wheelchair skills training: current practices in Canadian rehabilitation centers. Disabil Rehabil Assist Technol. 2015;10(5):393-400. doi: 10.3109/17483107.2014.907367. Epub 2014 Apr 7. PMID 24702608
- [Background] Gill TM, Baker DI, Gottschalk M, Peduzzi PN, Allore H, Byers A. A program to prevent functional decline in physically frail, elderly persons who live at home. N Engl J Med. 2002 Oct 3;347(14):1068-74. doi: 10.1056/NEJMoa020423. PMID 12362007
- [Background] Tousignant M, Dubuc N, Hebert R, Coulombe C. Home-care programmes for older adults with disabilities in Canada: how can we assess the adequacy of services provided compared with the needs of users? Health Soc Care Community. 2007 Jan;15(1):1-7. doi: 10.1111/j.1365-2524.2006.00645.x. PMID 17212620
- [Background] Sanford JA, Griffiths PC, Richardson P, Hargraves K, Butterfield T, Hoenig H. The effects of in-home rehabilitation on task self-efficacy in mobility-impaired adults: A randomized clinical trial. J Am Geriatr Soc. 2006 Nov;54(11):1641-8. doi: 10.1111/j.1532-5415.2006.00913.x. PMID 17087689
- [Background] Tousignant M, Boissy P, Corriveau H, Moffet H. In home telerehabilitation for older adults after discharge from an acute hospital or rehabilitation unit: A proof-of-concept study and costs estimation. Disabil Rehabil Assist Technol. 2006 Sep;1(4):209-16. doi: 10.1080/17483100600776965. PMID 19260168
- [Background] Lemay V, Routhier F, Noreau L, Phang SH, Ginis KA. Relationships between wheelchair skills, wheelchair mobility and level of injury in individuals with spinal cord injury. Spinal Cord. 2012 Jan;50(1):37-41. doi: 10.1038/sc.2011.98. Epub 2011 Sep 20. PMID 21931330
- [Background] Giesbrecht EM, Miller WC. Effect of an mHealth Wheelchair Skills Training Program for Older Adults: A Feasibility Randomized Controlled Trial. Arch Phys Med Rehabil. 2019 Nov;100(11):2159-2166. doi: 10.1016/j.apmr.2019.06.010. Epub 2019 Jul 20. PMID 31336101
- [Background] Sakakibara BM, Miller WC, Rushton PW. Rasch analyses of the wheelchair use confidence scale. Arch Phys Med Rehabil. 2015 Jun;96(6):1036-44. doi: 10.1016/j.apmr.2014.11.005. Epub 2014 Nov 25. PMID 25461823
- [Background] Kirby RL, Gillis DJ, Boudreau AL, Smith C, Rushton P, Clark-Gallant L, Parker KE, Webber A. Effect of a high-rolling-resistance training method on the success rate and time required to learn the wheelchair wheelie skill: a randomized controlled trial. Am J Phys Med Rehabil. 2008 Mar;87(3):204-11; quiz 212-4. doi: 10.1097/PHM.0b013e318164aa27. PMID 18287817
- [Background] Bratter B and Freeman E. The maturing of peer counselling. Generations 1990; 14: 49-52
- [Background] Bandura A. Self-efficacy: the exercise of control. New York: W. H. Freeman and Company, 1997.
- [Background] Ryan RM, Deci EL. Self-determination theory and the facilitation of intrinsic motivation, social development, and well-being. Am Psychol. 2000 Jan;55(1):68-78. doi: 10.1037//0003-066x.55.1.68. PMID 11392867
- [Background] Wilson P, Rodgers W, Blanchard C, et al. The relationship between psychological needs, self-determined motivation, exercise attitudes and physical fitness. Journal of Applied Social Psychology 2003; 33: 2373-2392.
- [Background] Atkinson M. eHealth in Canada: current trends and future challenges. Ottawa: Information and Communications Technology Council, 2009.
- [Background] Protheroe J, Blakeman T, Bower P, Chew-Graham C, Kennedy A. An intervention to promote patient participation and self-management in long term conditions: development and feasibility testing. BMC Health Serv Res. 2010 Jul 14;10:206. doi: 10.1186/1472-6963-10-206. PMID 20630053
- [Background] Ding D, Cooper RA and Pearlman J. Incorporating participatory action design into research and education. In: International Conference on Engineering Education Coimbra, Portugal, 2007.
- [Background] Giesbrecht EM, Miller WC, Mitchell IM, Woodgate RL. Development of a wheelchair skills home program for older adults using a participatory action design approach. Biomed Res Int. 2014;2014:172434. doi: 10.1155/2014/172434. Epub 2014 Sep 4. PMID 25276768
- [Background] Wild D, Grove A, Martin M, Eremenco S, McElroy S, Verjee-Lorenz A, Erikson P; ISPOR Task Force for Translation and Cultural Adaptation. Principles of Good Practice for the Translation and Cultural Adaptation Process for Patient-Reported Outcomes (PRO) Measures: report of the ISPOR Task Force for Translation and Cultural Adaptation. Value Health. 2005 Mar-Apr;8(2):94-104. doi: 10.1111/j.1524-4733.2005.04054.x. PMID 15804318
- [Background] Giesbrecht EM, Miller WC, Woodgate RL. Navigating uncharted territory: a qualitative study of the experience of transitioning to wheelchair use among older adults and their care providers. BMC Geriatr. 2015 Jul 28;15:91. doi: 10.1186/s12877-015-0092-2. PMID 26215495
- [Background] van den Berg-Emons RJ, Bussmann JB, Haisma JA, Sluis TA, van der Woude LH, Bergen MP, Stam HJ. A prospective study on physical activity levels after spinal cord injury during inpatient rehabilitation and the year after discharge. Arch Phys Med Rehabil. 2008 Nov;89(11):2094-101. doi: 10.1016/j.apmr.2008.04.024. PMID 18996237
- [Background] Page SJ, Persch AC. Recruitment, retention, and blinding in clinical trials. Am J Occup Ther. 2013 Mar-Apr;67(2):154-61. doi: 10.5014/ajot.2013.006197. PMID 23433269
- [Background] Sygna K, Johansen S, Ruland CM. Recruitment challenges in clinical research including cancer patients and their caregivers. A randomized controlled trial study and lessons learned. Trials. 2015 Sep 25;16:428. doi: 10.1186/s13063-015-0948-y. Erratum In: Trials. 2016 Mar 10;17(1):133. doi: 10.1186/s13063-016-1276-6. PMID 26407547
- [Background] Cook WL, Schiller C, McAllister MM, Hanson HM, Brasher PM, Donaldson MG, Macri E, Preto R, Guy P, Ashe MC. Feasibility of a follow-up hip fracture clinic. J Am Geriatr Soc. 2015 Mar;63(3):598-9. doi: 10.1111/jgs.13285. No abstract available. PMID 25800911
- [Background] Blanton S, Morris DM, Prettyman MG, McCulloch K, Redmond S, Light KE, Wolf SL. Lessons learned in participant recruitment and retention: the EXCITE trial. Phys Ther. 2006 Nov;86(11):1520-33. doi: 10.2522/ptj.20060091. PMID 17079752
- [Background] Gomes R, Michaelsen S, Rodrigues L, et al. Scientific research with individual post stroke: difficulties in recruitment, allocation and adherence on two different protocols of physiotherapy intervention. Fisioterapia e Pesquisa 2015; 22: 34-40. DOI: 10.590/1809-2950/13111022012015.
- [Background] McMurdo ME, Roberts H, Parker S, Wyatt N, May H, Goodman C, Jackson S, Gladman J, O'Mahony S, Ali K, Dickinson E, Edison P, Dyer C; Age and Ageing Specialty Group, NIHR, Comprehensive Clinical Research Network. Improving recruitment of older people to research through good practice. Age Ageing. 2011 Nov;40(6):659-65. doi: 10.1093/ageing/afr115. Epub 2011 Sep 11. PMID 21911335
- [Background] Best KL, Routhier F and Miller WC. Older adults' perceptions and experiences with a peer-led wheelchair training program. 34th International Seating Symposium. Vancouver, BC, 2018.
- [Background] Miller WC, Garden J, Mortenson WB. Measurement properties of the wheelchair outcome measure in individuals with spinal cord injury. Spinal Cord. 2011 Sep;49(9):995-1000. doi: 10.1038/sc.2011.45. Epub 2011 May 17. PMID 21577219
- [Background] Mortenson WB, Miller WC, Miller-Pogar J. Measuring wheelchair intervention outcomes: development of the wheelchair outcome measure. Disabil Rehabil Assist Technol. 2007 Sep;2(5):275-85. doi: 10.1080/17483100701475863. PMID 19263533
- [Background] Bowman J, Mogensen L, Marsland E, Lannin N. The development, content validity and inter-rater reliability of the SMART-Goal Evaluation Method: A standardised method for evaluating clinical goals. Aust Occup Ther J. 2015 Dec;62(6):420-7. doi: 10.1111/1440-1630.12218. Epub 2015 Aug 19. PMID 26286379
- [Background] Cress ME, Buchner DM, Prohaska T, Rimmer J, Brown M, Macera C, Dipietro L, Chodzko-Zajko W. Best practices for physical activity programs and behavior counseling in older adult populations. J Aging Phys Act. 2005 Jan;13(1):61-74. doi: 10.1123/japa.13.1.61. PMID 15677836
- [Background] World Health Organization. International classification of functioning disability and health. Geneva: World Health Organization, 2001.
- [Background] Talo C, Mannarini T and Rochira A. Sense of community and community participation: A meta-analytic review. Social Indicators Research 2014; 117: 1-28. DOI: 10.1007/s11205-013-0347-2.
- [Background] Kenny S and Gowran RJ. Outcome Measures for Wheelchair and Seating Provision: A Critical Appraisal. British Journal of Occupational Therapy 2014; 77: 67-77. DOI: 10.4276/030802214x13916969447119.
- [Background] Mortenson WB, Miller WC, Auger C. Issues for the selection of wheelchair-specific activity and participation outcome measures: a review. Arch Phys Med Rehabil. 2008 Jun;89(6):1177-86. doi: 10.1016/j.apmr.2008.01.010. PMID 18503817
- [Background] Auger C, Demers L, Gelinas I, Routhier F, Mortenson WB, Miller WC. Reliability and validity of the telephone administration of the wheelchair outcome measure (WhOM) for middle-aged and older users of power mobility devices. J Rehabil Med. 2010 Jun;42(6):574-81. doi: 10.2340/16501977-0557. PMID 20549163
- [Background] Fliess-Douer O, Vanlandewijck YC, Lubel Manor G, Van Der Woude LH. A systematic review of wheelchair skills tests for manual wheelchair users with a spinal cord injury: towards a standardized outcome measure. Clin Rehabil. 2010 Oct;24(10):867-86. doi: 10.1177/0269215510367981. Epub 2010 Jun 16. PMID 20554638
- [Background] Kilkens OJ, Post MW, Dallmeijer AJ, Seelen HA, van der Woude LH. Wheelchair skills tests: a systematic review. Clin Rehabil. 2003 Jul;17(4):418-30. doi: 10.1191/0269215503cr633oa. PMID 12785251
- [Background] Kirby RL, Dupuis DJ, Macphee AH, Coolen AL, Smith C, Best KL, Newton AM, Mountain AD, Macleod DA, Bonaparte JP. The wheelchair skills test (version 2.4): measurement properties. Arch Phys Med Rehabil. 2004 May;85(5):794-804. doi: 10.1016/j.apmr.2003.07.007. PMID 15129405
- [Background] Rushton PW, Kirby RL, Miller WC. Manual wheelchair skills: objective testing versus subjective questionnaire. Arch Phys Med Rehabil. 2012 Dec;93(12):2313-8. doi: 10.1016/j.apmr.2012.06.007. Epub 2012 Jun 21. PMID 22728701
- [Background] Rushton PW, Miller WC, Lee Kirby R, Eng JJ, Yip J. Development and content validation of the Wheelchair Use Confidence Scale: a mixed-methods study. Disabil Rehabil Assist Technol. 2011;6(1):57-66. doi: 10.3109/17483107.2010.512970. PMID 20809874
- [Background] Sakakibara BM, Miller WC, Eng JJ, Backman CL, Routhier F. Preliminary examination of the relation between participation and confidence in older manual wheelchair users. Arch Phys Med Rehabil. 2013 Apr;94(4):791-4. doi: 10.1016/j.apmr.2012.09.016. Epub 2012 Sep 27. PMID 23022451
- [Background] Berardi A, De Santis R, Tofani M, Marquez MA, Santilli V, Rushton PW, Mollica R, Galeoto G. The Wheelchair Use Confidence Scale: Italian translation, adaptation, and validation of the short form. Disabil Rehabil Assist Technol. 2018 Aug;13(6):575-580. doi: 10.1080/17483107.2017.1357053. Epub 2017 Jul 31. PMID 28758517
- [Background] Jones CA, Feeny D, Eng K. Test-retest reliability of health utilities index scores: evidence from hip fracture. Int J Technol Assess Health Care. 2005 Summer;21(3):393-8. doi: 10.1017/s0266462305050518. PMID 16110720
- [Background] Torrance GW, Furlong W, Feeny D. Health utility estimation. Expert Rev Pharmacoecon Outcomes Res. 2002 Apr;2(2):99-108. doi: 10.1586/14737167.2.2.99. PMID 19807322
- [Background] Luo N, Johnson J, Coons SJ. Using instrument-defined health state transitions to estimate minimally important differences for four preference-based health-related quality of life instruments. Med Care. 2010 Apr;48(4):365-71. doi: 10.1097/mlr.0b013e3181c162a2. PMID 20355266
- [Background] Sakakibara BM, Routhier F, Miller WC. Wheeled-mobility correlates of life-space and social participation in adult manual wheelchair users aged 50 and older. Disabil Rehabil Assist Technol. 2017 Aug;12(6):592-598. doi: 10.1080/17483107.2016.1198434. Epub 2016 Jul 4. PMID 27377171
- [Background] Sonenblum SE, Sprigle S, Caspall J, Lopez R. Validation of an accelerometer-based method to measure the use of manual wheelchairs. Med Eng Phys. 2012 Jul;34(6):781-6. doi: 10.1016/j.medengphy.2012.05.009. Epub 2012 Jun 12. PMID 22698978
- [Background] Sonenblum SE, Sprigle S, Lopez RA. Manual wheelchair use: bouts of mobility in everyday life. Rehabil Res Pract. 2012;2012:753165. doi: 10.1155/2012/753165. Epub 2012 Jul 15. PMID 22848837
- [Background] Tabachnick BG and Fidell LS. Using multivariate statistics. 5th ed. Boston: Pearson Education, 2007.
- [Background] Vickers AJ. Analysis of variance is easily misapplied in the analysis of randomized trials: a critique and discussion of alternative statistical approaches. Psychosom Med. 2005 Jul-Aug;67(4):652-5. doi: 10.1097/01.psy.0000172624.52957.a8. PMID 16046383
- [Background] Mbuagbaw L, Aves T, Shea B, Jull J, Welch V, Taljaard M, Yoganathan M, Greer-Smith R, Wells G, Tugwell P. Considerations and guidance in designing equity-relevant clinical trials. Int J Equity Health. 2017 Jun 5;16(1):93. doi: 10.1186/s12939-017-0591-1. PMID 28583125
- [Background] Brazier JE, Harper R, Jones NM, O'Cathain A, Thomas KJ, Usherwood T, Westlake L. Validating the SF-36 health survey questionnaire: new outcome measure for primary care. BMJ. 1992 Jul 18;305(6846):160-4. doi: 10.1136/bmj.305.6846.160. PMID 1285753
- [Background] Froehlich-Grobe K, Andresen EM, Caburnay C, White GW. Measuring health-related quality of life for persons with mobility impairments: an enabled version of the short-form 36 (SF-36E). Qual Life Res. 2008 Jun;17(5):751-70. doi: 10.1007/s11136-008-9342-5. Epub 2008 Apr 22. PMID 18427950
- [Derived] Giesbrecht E, Best KL, Miller WC, Routhier F, Harrison KL, Faieta J, Laberge M. Outcomes retention and impact of demographic characteristics and engagement for a community-based peer-led eHealth wheelchair skills training program. Disabil Rehabil Assist Technol. 2026 Feb 6:1-12. doi: 10.1080/17483107.2026.2623650. Online ahead of print. PMID 41649466
- [Derived] Giesbrecht E, Best KL, Miller WC, Routhier F, Harrison KL, Faieta J, Laberge M. Effect of a Community-Based Peer-Led eHealth Wheelchair Skills Training Program: A Randomized Control Trial. Arch Phys Med Rehabil. 2025 Jun;106(6):821-827. doi: 10.1016/j.apmr.2024.12.011. Epub 2024 Dec 19. PMID 39709023
- See also: Dalhousie University. Wheelchair Specifications Form — http://www.wheelchairskillsprogram.ca